CLINICAL TRIAL: NCT07010367
Title: Effects and Mechanism of Baliao Acupoint Stimulation (BL31~BL34) for Functional Constipation
Brief Title: Baliao Acupoint Stimulation toTreat Functional Constipation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Nanjing University of Chinese Medicine (Other)
Collaborators: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-056-SO
Record Dates: First submitted 2025-05-26; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Functional Constipation (FC)
Keywords: functional constipation; fMRI
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- acupuncture group (Experimental): Patients will receive acupuncture at Baliao acupuncts.
  Interventions: Procedure: Acupuncture
- sham group (Sham Comparator): Patients will receive sham acupuncture treatment.
  Interventions: Procedure: Sham acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Patients will be instructed to lie in the supine position. After strict disinfection of the acupoints area, acupuncture needles will be inserted into the Baliao points (inserted at the surface projections of the first, second, and third pairs of sacral foramina, with a depth of 3-4 cm). The treatment will be administered five times per week, with each session lasting 30 minutes, for a total of two weeks.
  Arms: acupuncture group
Procedure: Sham acupuncture — Patients will be instructed to lie in the supine position. After strict disinfection of the sham acupoints area, acupuncture needles will be inserted lateral to the surface projections of the first, second, and third pairs of sacral foramina, with a depth of 1 cm.The treatment will be administered five times per week, with each session lasting 30 minutes, for a total of two weeks.
  Arms: sham group

SUMMARY:
This study is a randomized controlled trial that explores how a specific acupuncture treatment might help people with functional constipation. The investigators are testing the idea that a treatment called "acupuncture at the Baliao acupoints" could work by changing the way certain parts of the brain connect and function. These brain changes might help improve gut function and relieve constipation symptoms.

The investigators will work with people who have functional constipation. Some participants will receive the real Baliao acupoint thread embedding, while others will get a sham acupuncture as a comparison. Using special brain imaging techniques, the investigators will look at how the brain's connections and structures change. The investigators will also track how often participants have bowel movements, the consistency of their stools, and their overall symptoms and quality of life. By comparing these results, the investigators hope to understand how the Baliao acupoint treatment works and why it might be effective for constipation.

ELIGIBILITY:
Inclusion Criteria:

* Age:18 years or older.
* Diagnosed with functional constipation according to the Rome IV criteria.
* The participant has not received any treatment for functional constipation in the past two weeks (except for emergency interventions).
* Right-handed.
* Signed a written informed consent form to participate in this study.

Exclusion Criteria:

* Presence of organic constipation, drug-induced constipation, or systemic constipation.
* Presence of metallic foreign bodies in the body, pacemakers, or other contraindications for MRI examination.
* Communication disorders or unwillingness to cooperate with treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-06-20 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Spontaneous bowel movements | SBMs will be recorded 1 week before treatment and at 2, 4, 6, and 8 weeks after treatment.
  Spontaneous bowel movements (SBMs) refers to the frequency of bowel movements that occur without the use of any medications or other aids within the past 24 hours. These data are collected from the constipation diaries filled out daily by patients with functional constipation (FC) to determine the weekly count of SBMs. The data collection time points include before treatment and at 2, 4, 6, and 8 weeks after treatment.

SECONDARY OUTCOMES:
PAC-SYM | PAC-SYM will be assessed at 1 week before treatment and at 2, 4, 6, and 8 weeks after treatment
  Patient Assessment of Constipation symptom(PAC-SYM) is a tool used to evaluate the symptoms and severity of constipation in patients. The scale consists of three sections: stool symptoms, rectal symptoms, and abdominal symptoms, with a total of 12 items. The score ranges from 0 to 48, with higher scores indicating more severe constipation symptoms.
PAC-QOL | PAC-QOL will be accessed 1 week before treatment and at 2, 4, 6, and 8 weeks after treatment.
  Patient Assessment of Constipation quality of life is a tool used to assess the impact of constipation on patients' quality of life. The scale, known as PAC-QOL, consists of four dimensions: Physical Discomfort (4 items), Psychosocial Discomfort (8 items), Worries and Discomfort (11 items), and Treatment Satisfaction (5 items), with a total of 28 items. The score ranges from 0 to 112, with higher scores indicating a greater negative impact of constipation on quality of life.

OTHER OUTCOMES:
SAS | SAS will be accessed 1 week before treatment and at 2, 4, 6, and 8 weeks after treatment.
  The Self-Rating Anxiety Scale (SAS) consists of 20 items that reflect subjective feelings of anxiety. Each item is rated on a four-point scale based on the frequency of symptom occurrence. Among these items, 15 are scored in the positive direction, while 5 are scored in the reverse direction. According to the Chinese normative data, the cutoff score for the standardized SAS score is 50. Scores ranging from 50 to 59 indicate mild anxiety, 60 to 69 indicate moderate anxiety, and scores above 69 indicate severe anxiety.
SDS | SDS will be accessed 1 week before treatment and at 2, 4, 6, and 8 weeks after treatment.
  Self-Rating Depression Scale (SDS) consists of 20 items that reflect subjective feelings of depression. Each item is rated on a four-point scale based on the frequency of symptom occurrence. Among these items, 10 are scored in the positive direction, and 10 are scored in the reverse direction. According to the Chinese normative data, the cutoff score for the standardized SDS score is 53. Scores ranging from 53 to 62 indicate mild depression, 63 to 72 indicate moderate depression, and scores above 72 indicate severe depression.
Amplitude of Low-Frequency Fluctuations | at 1 week before treatment and 4 weeks after treatment
  Amplitude of Low-Frequency Fluctuations(ALFF) is a common used measurement when analyzing functional MRI. iIt calculates the low-frequency amplitude values of each voxel to observe the magnitude of changes in blood oxygen level-dependent (BOLD) signals relative to the baseline. It can sensitively reflect abnormal activities in the regions of interest in the brain.

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data contains highly sensitive and personal information about study participants. Sharing IPD could potentially compromise participant privacy and confidentiality.